CLINICAL TRIAL: NCT00806741
Title: Role of Nitric Oxide in Optic Nerve Head Blood Flow Regulation During Isometric Exercise in Healthy Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Assoc. Prof. PD Dr., Medical University of Vienna
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: OPHT-300708
Record Dates: First submitted 2008-12-10; First posted 2008-12-11 (Estimated); Last update posted 2012-11-30 (Estimated); Status verified 2012-11

CONDITIONS: Healthy
Keywords: L-NG-Monomethyl Arginine; Optic Nerve Head blood flow; Intraocular Pressure; Regional blood flow; Ocular Physiology; Optic Disk
MeSH Terms: interventions — omega-N-Methylarginine; Phenylephrine; Laser-Doppler Flowmetry

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): NG-monomethyl-L-arginine (L-NMMA)
  Interventions: Drug: NG-monomethyl-L-arginine (L-NMMA); Device: Laser Doppler Flowmetry; Device: Goldmann applanation tonometer; Other: squatting
- 2 (Active Comparator): Phenylephrine
  Interventions: Drug: Phenylephrine; Device: Laser Doppler Flowmetry; Device: Goldmann applanation tonometer; Other: squatting
- 3 (Placebo Comparator): Physiological saline solution
  Interventions: Drug: Physiological saline solution (as placebo); Device: Laser Doppler Flowmetry; Device: Goldmann applanation tonometer; Other: squatting

INTERVENTIONS:
Drug: NG-monomethyl-L-arginine (L-NMMA) — bolus 6mg/kg over 5 minutes followed by a continuous infusion of 60µg/kg/min over 15 minutes
  Arms: 1
Drug: Phenylephrine — 1μg/kg/min, infusion period 20 minutes
  Arms: 2
Drug: Physiological saline solution (as placebo) — infusion period 20 minutes
  Arms: 3
Device: Laser Doppler Flowmetry — blood flow measurements at the temporal neuroretinal rim of the optic nerve head
Device: Goldmann applanation tonometer — intraocular pressure measurements
Other: squatting — Subjects will perform squatting for 6 minutes while blood flow is measured

SUMMARY:
Autoregulation is defined as the ability of a vascular bed to adapt its vascular resistance to changes in perfusion pressure. In the eye, several studies have reported that retinal blood flow is autoregulated over a wide range of ocular perfusion pressures. The investigators recently showed that nitric oxide (NO) is a key metabolite in the regulation of vascular tone in the eye and plays an important role in the blood flow autoregulation of the choroidal circulation. However, no data is yet available for the optic nerve head. Thus, the present study is designed to test the hypothesis that NO plays also a role in optic nerve head blood flow autoregulation. Therefore, subjects will perform squatting to increase systemic perfusion pressure during administration of either a nitric oxide synthase inhibitor (L-NMMA), an α-receptor agonist (phenylephrine) or placebo. Optic nerve head blood flow will be continuously measured during the procedure to investigate optic nerve head autoregulation.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 18 and 35 years, nonsmokers
* Men and women will be included in equal parts
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant
* Normal findings in the laboratory testings unless the investigator considers an abnormality to be clinically irrelevant
* Normal ophthalmic findings, ametropia less than 3 diopters

Exclusion Criteria:

* Regular use of medication, abuse of alcoholic beverages, participation in a clinical trial in the 3 weeks preceding the study
* Treatment in the previous 3 weeks with any drug (except intake of oral contraceptives)
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* History or presence of gastrointestinal, liver or kidney disease, or other conditions known to interfere with distribution, metabolism or excretion of study drugs
* Blood donation during the previous 3 weeks
* Pregnancy

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2009-09; Primary Completion 2010-03 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Optic nerve head pressure-flow relationship | in total 6x on 3 study days

CONTACTS AND LOCATIONS:
Overall Officials: Gabriele Fuchsjaeger-Mayrl, MD, Univ.Doz., Principal Investigator — Medical University of Vienna
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Derived] Schmidl D, Boltz A, Kaya S, Lasta M, Pemp B, Fuchsjager-Mayrl G, Hommer A, Garhofer G, Schmetterer L. Role of nitric oxide in optic nerve head blood flow regulation during isometric exercise in healthy humans. Invest Ophthalmol Vis Sci. 2013 Mar 15;54(3):1964-70. doi: 10.1167/iovs.12-11406. PMID 23439596